CLINICAL TRIAL: NCT00658203
Title: Clinical Evaluation on Advanced Resynchronization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: P. RITTER - Principal investigator, InParys
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLEAR - IPEA01
Record Dates: First submitted 2008-03-28; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: CRT-P; PEA; Severe Heart Failure (NYHA Class III or IV); Cardiomyopathy of any etiology; Sinus rhythm; Reduced Left-Ventricular Ejection Fraction; LVEDD>30 mm/m2; QRS Duration: > 150 ms or > 120 ms; Aortic Pre-Ejection Delay > 140 ms; Interventricular Mechanical Delay > 40 ms; Delayed activation of postero-lateral Left Ventricular wall; Optimal and stable pharmacological treatment
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): PEA optimized CRT
  Interventions: Device: New Living CHF
- 2 (Other): Standard optimized CRT
  Interventions: Device: New Living CHF

INTERVENTIONS:
Device: New Living CHF — PEA CRT optimization
  Arms: 1
Device: New Living CHF — Standard optimized CRT.
  Arms: 2

SUMMARY:
The aim of the study is to compare clinical benefits of the cardiac resynchronisation (CRT) achieved by the PEA optimised pacing configuration and a CRT optimised by standard clinical procedure.

PEA optimised configuration (PEA-CRT) is obtained, during patient's follow-up, using the Peak Endocardial Acceleration sensor features onboard the device.

DETAILED DESCRIPTION:
The study is a prospective, multicentre, controlled and randomised clinical investigation, with two single-blinded arms.

The objective of the study is to compare the clinical benefits of Cardiac Resynchronisation Therapy (CRT) optimised by automatic PEA sensor features (PEA-CRT), with those obtained by standard optimisation procedure (STD-CRT).

The patient candidate for inclusion in the study has a severe chronic Heart Failure, indicated for the implantation of a Biventricular pacing system according to updated ESC guidelines (2005).

All patients included in the study will be followed-up for 1 year; patient's follow-ups are scheduled during hospitalisation, at one month, 3 months, 6 months and one year after implantation.

ELIGIBILITY:
Inclusion Criteria:

The patient candidate for inclusion in the study must be indicated for implantation of a Biventricular pacing system, with the following clinical conditions:

* Severe Heart Failure (NYHA Class III or IV)
* Cardiomyopathy of any etiology
* Sinus rhythm
* Reduced Left-Ventricular Ejection Fraction
* Left-Ventricular End Diastolic Diameter greater than or equal to 30 mm/m2 (LVEDD>30 mm/m2)
* QRS Duration:

  * > 150 ms or
  * > 120 ms and documented Mechanical Dissynchrony (by ECHO) meeting two out of three of the following criteria:

    * Aortic Pre-Ejection Delay > 140 ms
    * Interventricular Mechanical Delay > 40 ms
    * Delayed activation of postero-lateral Left Ventricular wall (after mitral valve opening)
* Optimal and stable (1 month before inclusion) pharmacological treatment, including, if tolerated, Beta Blockers, Angiotensin-Converting Enzyme (ACE) Inhibitors or ACE Inhibitor substitutes, Spironolactone, and diuretics

Exclusion Criteria:

Any patient who has one of the following characteristics will be excluded from the study:

* ICD indication (Life-threatening ventricular arrhythmias)
* Persistent or permanent Atrial Arrhythmia without possibility to restore sinus rhythm (spontaneous termination, anti-tachycardia pacing, pharmacological or electrical cardioversion).
* Patient already implanted with a conventional pacemaker device
* Myocardial infarction within the last three months
* Heart surgery, or revascularization within the last three months, or expected
* Heart surgery refused because of co-morbidity factors
* Included in transplantation list
* Already enrolled in other study
* Life expectancy less than 1 year
* Pregnancy
* Age less than 18
* Forfeiture of freedom or under guardianship
* Not able to understand the aim of the study and its procedures
* Refusing to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be evaluated at 1 year (M12), in term of improved, unchanged or worsened patient's conditions, with a composite analysis of NYHA class evolution, heart-failure-related hospitalisations and Quality of Life evaluation. | 12 months

SECONDARY OUTCOMES:
PEA-CRT optimisation is at least effective as the standard optimisation in term of efficacy of the therapy and patients' quality of life. | 12 months
PEA is an index of the patients' clinical status and allows to predict acute HF episode in both arms. | 12 months
Efficacy of the therapy comparing the two arms in terms of NYHA | 12 months
Efficacy of the therapy comparing the two arms in terms of Cardiovascular mortality | 12 months
Efficacy of the therapy comparing the two arms in terms of Heart Failure Quality Of Life (EuroQoL-5D) score | 12 months
Efficacy of the therapy comparing the two arms in terms of BNP dosage | 12 months
Efficacy of the therapy comparing the two arms in terms of Number and duration of heart-failure-related patient's hospitalisations, during the study period. | 12 months
Efficacy of the therapy comparing the two arms in terms of Left Ventricular End Diastolic Diameter | 12 months
Efficacy of the therapy comparing the two arms in terms of Left Ventricular End Systolic Diameter | 12 months
Efficacy of the therapy comparing the two arms in terms of Left Ventricular Ejection Fraction | 12 months
Efficacy of the therapy comparing the two arms in terms of Left Pre-Ejection Interval | 12 months
Efficacy of the therapy comparing the two arms in terms of Right Pre-Ejection Interval | 12 months
Efficacy of the therapy comparing the two arms in terms of Total Duration of Left Systole | 12 months
Efficacy of the therapy comparing the two arms in terms of E velocity | 12 months
Efficacy of the therapy comparing the two arms in terms of A velocity | 12 months
Efficacy of the therapy comparing the two arms in terms of Ventricular spike-Mitral valve closure interval | 12 months
Efficacy of the therapy comparing the two arms in terms of Ventricular spike-Mitral valve opening interval | 12 months
Efficacy of the therapy comparing the two arms in terms of Mitral Valve regurgitation. | 12 months
Time spent to achieve the CRT optimal configuration during each follow-up | 12 months
PEA monitoring and prognostic relevance correlating the PEA diagnostic trends with the parameters used to asses the efficacy of the therapy and patients' quality of life (NYHA class, mortality, HF-hospitalisation, EuroQoL-5D score, BNP dosage, Echo | 12 months
(LVEF) comparing the changes Left Ventricular Ejection Fraction in the two arms with an intermediate analysis at 6 months done by a Core Centre. | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: P Ritter, Dr, Principal Investigator — InParys Cardiologie
Locations (36):
- France (12):
  - CH Albi, Albi
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CH Lomme, Lomme
  - CHU Montpellier, Montpellier
  - NC Nantaises, Nantes
  - CH Pau, Pau
  - CHU Poitiers, Poitiers
  - CHR Cardiologie A, Rennes
  - CHU Rouen, Rouen
  - CH Yves le Foll, Saint-Brieuc
  - InParys Cardiology, Saint-Cloud
- Germany (4):
  - UKB Unfallkrankenhaus, Berlin
  - Univ Saarland, Homburg
  - Stiftsklinikum Augustinum, München
  - St.Adolfstift, Reinbek
- Italy (7):
  - Osp. B. Ramazzini, Carpi
  - Osp. Civile, Desio
  - Osp. S. Maria Nuova, Florence
  - Osp. Univ. Careggi, Florence
  - Osp. Niguarda, Milan
  - Osp. Civile, Rieti
  - Osp. S. Filippo Neri, Rome
- Netherlands (4):
  - Medisch Centrum Rijnmond-Zuid, Rotterdam
  - Diaconessenhuis, Utrecht
  - Vlietland Ziekenhuis, Vlaardingen
  - Isala Klinieken, Zwolle
- Spain (4):
  - H. General Universit., Alicante
  - H. Virgen de las Nieves, Granada
  - H. General Universit., Valencia
  - Hosp. Clinico, Valencia
- United Kingdom (5):
  - Royal Hospital, Bournemouth
  - Saint Peter's Hospital, Chertsey
  - General Hospital, Eastbourne
  - Nothern General, Sheffield
  - University Hospital, Southampton